CLINICAL TRIAL: NCT00084669
Title: Targeting Insomnia to Enhance Hot Flush Treatment in Women Receiving Therapy for Breast Cancer or Breast Cancer Risk-Reduction
Brief Title: Venlafaxine With or Without Zolpidem in Treating Hot Flashes and Associated Sleep Disorders in Women With Breast Cancer OR at High Risk for Developing Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Hadine Joffe, MD, Massachusetts General Hospital
Allocation: Randomized | Masking: Double | Purpose: Supportive Care
Other Study IDs: CDR0000365502; MGH-DFCI-02311; DFCI-02311
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: Breast Cancer; Hot Flashes; Sleep Disorders
Keywords: hot flashes; sleep disorders; ductal breast carcinoma in situ; breast cancer in situ; lobular breast carcinoma in situ; lobular breast carcinoma; recurrent breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms; Hot Flashes; Sleep Wake Disorders; Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ; Carcinoma, Lobular | interventions — Venlafaxine Hydrochloride; Zolpidem

INTERVENTIONS:
Drug: venlafaxine
Drug: zolpidem tartrate
Procedure: management of therapy complications

SUMMARY:
RATIONALE: Venlafaxine may be effective in relieving hot flashes caused by hormone therapy. Giving venlafaxine with zolpidem (a sleeping pill) may improve sleep and quality of life in women who are receiving hormone therapy for treatment or prevention of breast cancer.

PURPOSE: This randomized clinical trial is studying giving venlafaxine together with zolpidem to see how well it works compared to venlafaxine alone in relieving hot flashes and associated sleep disorders in women who are receiving hormone therapy to treat or prevent breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effect of venlafaxine or another serotonin-reuptake inhibitor with vs without zolpidem, in terms of sleep continuity, in women with breast cancer or at high risk for developing breast cancer who experience hot flushes and associated sleep disorders.
* Compare quality of life in patients treated with these regimens.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients are stratified by concurrent use of serotonin-reuptake inhibitors (SRI).

* Stratum 1 (no concurrent SRI): Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive oral venlafaxine once daily and oral zolpidem once daily for 5 weeks*.
  * Arm II: Patients receive oral venlafaxine once daily and oral placebo once daily for 5 weeks*.
* Stratum 2 (concurrently on SRI): Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive oral zolpidem once daily for 5 weeks*.
  * Arm II: Patients receive oral placebo once daily for 5 weeks*. NOTE: *After 5 weeks of study treatment, patients in stratum 1 may taper or continue venlafaxine over 2 weeks (for a total duration of venlafaxine use of 7 weeks); patients in arm I of both strata may taper or continue zolpidem over 1 week (for a total duration of zolpidem use of 6 weeks); continuation or tapering of drugs in both arms occurs in an open-label fashion off study.

In both strata, treatment continues in the absence of unacceptable toxicity.

In both strata, hot flushes, sleep continuity, sleep quality, and quality of life are assessed at baseline and at weeks 1, 3, and 6.

PROJECTED ACCRUAL: A total of 119 patients will be accrued for this study within 20 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* At increased risk of developing breast cancer, meeting 1 of the following criteria:

  * Diagnosis of 1 of the following:

    * Ductal carcinoma in situ
    * Invasive breast cancer
    * Lobular carcinoma in situ
    * Atypical ductal or lobular hyperplasia
    * Lobular carcinoma
  * Candidate for breast cancer risk reduction for any of the following:

    * Predisposing mutation in a breast cancer susceptibility gene
    * Prior chest radiotherapy for Hodgkin's disease
    * Gail model score > 1.67% over 5 years
* Experiencing daytime and nocturnal hot flushes at least 14 times per week within the past 2 weeks
* Experiencing sleep disturbance, characterized by the presence of all of the following for ≥ 1 month:

  * ≥ 3 awakenings per night occurring ≥ 3 nights per week
  * Insomnia impedes daytime function
  * Hot flushes are the primary cause of insomnia (determined at baseline visit)
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 to 65

Sex

* Female

Menopausal status

* Not specified

Performance status

* ECOG 0-1

Life expectancy

* At least 6 months

Hematopoietic

* Not specified

Hepatic

* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN

Renal

* Creatinine ≤ 1.5 times ULN

Cardiovascular

* No clinically significant cardiac disease
* No uncontrolled hypertension within the past 3 months, defined as the following:

  * Diastolic blood pressure > 95 mm Hg on > 1 occasion
  * Systolic blood pressure > 160 mm Hg on > 1 occasion

Pulmonary

* No clinically significant respiratory disease

Psychiatric

* Beck depression inventory score ≤ 15
* No active panic or depressive disorder within the past month
* No lifetime history of bipolar or psychotic disorder
* No active substance-use disorders, including alcohol and benzodiazepines, within the past year
* No suicidal or homicidal ideation
* No hypomania or mania

Other

* No prior adverse reaction to venlafaxine or zolpidem
* None of the following sleep disorders within the past 6 months:

  * Sleep apnea
  * Narcolepsy
  * Periodic limb movement disturbance
* No abuse or misuse of study medication
* No daytime sedation that interferes with ability to function
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 1 month after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* More than 3 months since prior chemotherapy
* No concurrent chemotherapy

Endocrine therapy

* More than 1 month since prior regular use (> 25% of the time) of oral, transdermal, or injection preparations of androgens, estrogens, or progestins

  * Vaginal suppositories and creams allowed
* No concurrent regular use of oral, transdermal, or injection preparations of androgens, estrogens, or progestins

Radiotherapy

* See Disease Characteristics
* More than 3 months since prior radiotherapy
* No concurrent radiotherapy

Surgery

* See Disease Characteristics

Other

* More than 1 month since prior regular use (> 25% of the time) of any of the following:

  * Hypnotic agents (e.g., benzodiazepines, zolpidem, zaleplon, trazodone, or diphenhydramine)
  * Clonidine
* More than 1 month since prior antidepressants or other medications that are known to influence mood > 25% of the time (no serotonin-reuptake inhibitors [SRI] stratum only)
* Concurrent SRI required provided they were initiated ≥ 1 month ago at or above the minimum dose, including any of the following (concurrent SRI stratum only):

  * Fluoxetine
  * Paroxetine
  * Paroxetine CR
  * Sertraline
  * Citalopram
  * S-citalopram
  * Venlafaxine
  * Fluvoxamine
* No concurrent warfarin
* No concurrent hypnotic agents, clonidine, or antidepressants, or other medications known to influence sleep, or mood

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Estimated)
Dates: Start 2004-05; Primary Completion 2007-10 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Sleep improvement by biologic data and actigraphy data at the end of study treatment

SECONDARY OUTCOMES:
Quality of life by BDI, QOLI, PSI, NCCTG symptom diary, PSQI, MOS SF-36 at the end of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hadine Joffe, MD, MSC, Study Chair — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts